CLINICAL TRIAL: NCT06121336
Title: PRecisiOn Medicine In StrokE Study on the Evolution of Plasma Brain-Derived Tau in 100 Patients With Acute Ischemic Stroke
Brief Title: PRecisiOn Medicine In StrokE: Evolution of Plasma Brain-Derived Tau in Acute Stroke
Acronym: PROMISE-BD-100
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Steffen Tiedt, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU_ISD_2023_PROMISE-BD-100
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Brain Ischemia; Nervous System Diseases
Keywords: Stroke; Brain injury; Biomarker; Pathophysiology
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Brain Ischemia; Nervous System Diseases; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic Stroke: 100 patients admitted to a specialized stroke service because of an acute ischemic stroke due to large- or medium-vessel occlusion within 9 hours of stroke onset. BD-tau levels and other suggested markers of brain injury (e.g.. NfL) will be assessed every hour from admission to 48 hours after onset. Routinely collected clinical data including from neuroimaging will be collected throughout hospitalization. Clinical follow-up will be performed at 3 months.
  Interventions: Diagnostic Test: Plasma levels of BD-tau

INTERVENTIONS:
Diagnostic Test: Plasma levels of BD-tau — Plasma levels of BD-tau will be assessed using a single-molecule array assay.

SUMMARY:
The investigators recently identified Brain-derived tau (BD-tau) as a sensitive blood-based biomarker for brain injury in acute ischemic stroke: in patients with acute ischemic stroke, plasma BD-tau was associated with imaging-based metrics of brain injury upon admission, increased within the first 24 hours in correlation with infarct progression, and at 24 hours was superior to final infarct volume in predicting 90-day functional outcome. While informing on the relation of BD-tau with imaging-based metrics of brain injury, this cross-sectional study was restricted to BD-tau assessments upon admission and at day 2 and could not inform on key characteristics of the evolution of plasma BD-tau, including when exactly it starts to rise, how long it continues to rise, and how it is determined by infarct characteristics as well as comorbidities. Here, the investigators aim to assess plasma BD-tau every hour from admission to 48 hours after onset to evaluate the hypothesis that BD-tau rises immediately after onset and plateaus between three and 48 hours after onset.

DETAILED DESCRIPTION:
Ischemic stroke remains a leading cause of death and long-term disability worldwide,1 despite major advancements in reperfusion therapies.2,3 While neuroimaging modalities have expanded patient eligibility for reperfusion therapies by estimating ischemic core and salvageable tissue,4-7 their assessments are mostly single-timed. Currently available clinical algorithms lack the capacity to continuously track the dynamic evolution of how the primary core progresses to a final infarct, which, however, is a major determinant of functional outcome.8-10 Monitoring infarct trajectories could support therapeutic decision-making in patients with large-vessel occlusion stroke and unveil determinants of stroke progression, aiding in patient selection for trials evaluating cytoprotection11 and targeting clinically ineffective reperfusion.12 Previously studied blood-based biomarkers such as Neurofilament Light Chain (NfL),13 neuron-specific enolase (NSE),14 glial fibrillary acidic protein (GFAP),15,16 and S 100 calcium-binding protein B (S100B)17 either failed to capture the extent of brain injury within the acute phase of stroke or lack specificity. Plasma levels of brain-derived tau (BD-tau) were recently found to show high value for monitoring brain injury in patients with acute ischemic stroke: In 502 patients with acute IS, plasma BD-tau was associated with imaging-based metrics of brain injury upon admission, increased within the first 24 hours in correlation with infarct progression, and at 24 hours was superior to final infarct volume in predicting 90-day functional outcome.18 While informing on the relation of BD-tau with imaging-based metrics of brain injury, this large cross-sectional study was restricted to BD-tau assessments upon admission (median time from onset: 4.4 hours) and at day 2 (median time from onset: 22.7 hours) and could not inform on key characteristics of the evolution of plasma BD-tau, including when exactly it starts to rise, how long it continues to rise, and how it is determined by infarct characteristics as well as comorbidities. That knowledge would be of great value to determine the responsiveness of plasma BD-tau to brain injury after onset and to evaluate whether BD-tau plateaus at different time points after onset indicating no further infarct progression. Here, the investigators hypothesize that BD-tau rises immediately after onset and plateaus between three and 48 hours after onset. PROMISE-BD-100 will thus assess BD-tau levels every hour from admission to 48 hours from stroke onset in patients that present with the clinical diagnosis of an acute ischemic stroke due to a large- or medium-vessel occlusion within 9 hours from symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute ischemic stroke
* presentation within 9 hours of symptom onset
* large- or medium-vessel occlusion (i.e. an occlusion of the ICA, MCA [segments M1-M4], ACA [segments A1-A3], basilar artery, or PCA [segments P1 to P3]) confirmed by CT or MRI angiography
* at least 18 years of age
* written informed consent

Exclusion Criteria:

* CT or MRI showing intracranial hemorrhage upon admission
* A history of ischemic stroke, subarachnoid hemorrhage, intracerebral hemorrhage, subdural hematoma, epidural hematoma, CNS tumor, meningitis, or encephalitis within the last three months
* severe renal dysfunction (eGFR < 30ml/min/1.73m2)
* dementia
* pre-stroke disability defined as a premorbid modified Rankin Scale score > 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited upon admission to a tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome are plasma BD-tau levels in acute ischemic stroke. | Every hour from admission to 48 hours after onset.
  The evolution of BD-tau levels will be characterized by:
  * the time point when plasma BD-tau levels start to rise after onset (defined as the earliest time point [in relation to onset] that showed higher BD-tau levels compared with the previous assessment and lower levels compared with the next assessment),
  * the type of rise (e.g. linear, exponential, or logarithmic), and
  * until when plasma BD-tau levels continue to rise (defined as the time point [in relation to onset] compared to which BD-tau levels do not increase by ≥ 5 % compared to 1h, 2h, and 3h afterwards). 5 % were chosen without prior knowledge and in an attempt to account for assay-dependent variations of BD-tau quantifications (coefficient of variation 8-9 %)18 while keeping a biologically and clinically plausible value (rather than e.g. 10 %).

SECONDARY OUTCOMES:
ASPECTS on non-contrast CT | Upon admission
Ischemic core volume on CT perfusion | Upon admission
Regional leptomeningeal collateral score on CT angiography | Upon admission
Final infarct volume | Between 48 hours after symptom onset and discharge (latest 10 days after onset)
  Final infarct volume will be assessed on delayed neuroimaging (CT or MRI), at least 48 after symptom onset.
Infarct progression | Between admission and discharge (latest 10 days after onset)
  Infarct progression is defined as the difference between ischemic core volume quantified on admission CT perfusion scans and infarct volume quantified on delayed neuroimaging.
90-day functional outcome | 90 days (± 14 days) after onset
  Functional outcome at 90 days (± 14 days) will be assessed using the modified Rankin Scale (mRS). The mRS is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
7-day functional outcome | 7 days after onset
  Functional outcome at 7 days (or discharge if earlier) will be assessed using the modified Rankin Scale (mRS). The mRS is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
Early recurrent ischemic stroke | Between admission and discharge (latest 10 days after onset)
  The diagnosis of an early recurrent ischemic stroke will be based on i) sudden onset of a new focal neurological deficit within the first seven days after the index stroke that can not be explained by other non-ischemic causes such as seizure, metabolic derangement, or other systemic conditions, and ii) the presence of a new DWI-positive lesion on MRI or a new ischemic lesion on a delayed CT scan that is distinct from the index stroke lesion and that is consistent with the new clinical symptoms.
Secondary intracerebral hemorrhage | Between admission and discharge (latest 10 days after onset)
  Secondary intracerebral hemorrhage is defined as a new intracerebral hemorrhage independent of the primary ischemic lesion that is observed between the initial hemorrhage-free neuroimaging scan and discharge
Hemorrhagic transformation | Between admission and discharge (latest 10 days after onset)
  The occurrence of hemorrhagic transformation will be evaluated based on the morphological ECASS criteria.20

OTHER OUTCOMES:
Plasma levels of NfL | Hourly from admission to 48 hours after onset
  Plasma levels of NfL will be assessed at an hourly basis using a single-molecule array assay.
Plasma levels of GFAP | Hourly from admission to 48 hours after onset
  Plasma levels of GFAP will be assessed at an hourly basis using a single-molecule array assay.
Plasma proteome and metabolome composition | Hourly from admission to 48 hours after onset
  Plasma proteome and metabolome composition will be assessed using mass spectrometry or alternatives.

CONTACTS AND LOCATIONS:
Locations (1):
- LMU University hospital, LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data, including data dictionaries, that underlie results in a publication, will be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and additional supporting information will become available starting 6 months after publication.
Access Criteria: IPD and additional supporting information will be shared with academic researchers with a reasonable request to the corresponding author of the respective publication.

REFERENCES:
- [Background] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721
- [Background] Thomalla G, Boutitie F, Ma H, Koga M, Ringleb P, Schwamm LH, Wu O, Bendszus M, Bladin CF, Campbell BCV, Cheng B, Churilov L, Ebinger M, Endres M, Fiebach JB, Fukuda-Doi M, Inoue M, Kleinig TJ, Latour LL, Lemmens R, Levi CR, Leys D, Miwa K, Molina CA, Muir KW, Nighoghossian N, Parsons MW, Pedraza S, Schellinger PD, Schwab S, Simonsen CZ, Song SS, Thijs V, Toni D, Hsu CY, Wahlgren N, Yamamoto H, Yassi N, Yoshimura S, Warach S, Hacke W, Toyoda K, Donnan GA, Davis SM, Gerloff C; Evaluation of unknown Onset Stroke thrombolysis trials (EOS) investigators. Intravenous alteplase for stroke with unknown time of onset guided by advanced imaging: systematic review and meta-analysis of individual patient data. Lancet. 2020 Nov 14;396(10262):1574-1584. doi: 10.1016/S0140-6736(20)32163-2. Epub 2020 Nov 8. PMID 33176180
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Turc G, Tsivgoulis G, Audebert HJ, Boogaarts H, Bhogal P, De Marchis GM, Fonseca AC, Khatri P, Mazighi M, Perez de la Ossa N, Schellinger PD, Strbian D, Toni D, White P, Whiteley W, Zini A, van Zwam W, Fiehler J. European Stroke Organisation - European Society for Minimally Invasive Neurological Therapy expedited recommendation on indication for intravenous thrombolysis before mechanical thrombectomy in patients with acute ischaemic stroke and anterior circulation large vessel occlusion. Eur Stroke J. 2022 Mar;7(1):I-XXVI. doi: 10.1177/23969873221076968. Epub 2022 Feb 17. PMID 35300256
- [Background] Turc G, Bhogal P, Fischer U, Khatri P, Lobotesis K, Mazighi M, Schellinger PD, Toni D, de Vries J, White P, Fiehler J. European Stroke Organisation (ESO) - European Society for Minimally Invasive Neurological Therapy (ESMINT) Guidelines on Mechanical Thrombectomy in Acute Ischaemic StrokeEndorsed by Stroke Alliance for Europe (SAFE). Eur Stroke J. 2019 Mar;4(1):6-12. doi: 10.1177/2396987319832140. Epub 2019 Feb 26. PMID 31165090
- [Background] Berge E, Whiteley W, Audebert H, De Marchis GM, Fonseca AC, Padiglioni C, de la Ossa NP, Strbian D, Tsivgoulis G, Turc G. European Stroke Organisation (ESO) guidelines on intravenous thrombolysis for acute ischaemic stroke. Eur Stroke J. 2021 Mar;6(1):I-LXII. doi: 10.1177/2396987321989865. Epub 2021 Feb 19. PMID 33817340
- [Background] Boulouis G, Lauer A, Siddiqui AK, Charidimou A, Regenhardt RW, Viswanathan A, Rost N, Leslie-Mazwi TM, Schwamm LH. Clinical Imaging Factors Associated With Infarct Progression in Patients With Ischemic Stroke During Transfer for Mechanical Thrombectomy. JAMA Neurol. 2017 Nov 1;74(11):1361-1367. doi: 10.1001/jamaneurol.2017.2149. PMID 28973081
- [Background] Ospel JM, McDonough R, Demchuk AM, Menon BK, Almekhlafi MA, Nogueira RG, McTaggart RA, Poppe AY, Buck BH, Roy D, Haussen DC, Chapot R, Field TS, Jayaraman MV, Tymianski M, Hill MD, Goyal M; ESCAPE-NA1 investigators. Predictors and clinical impact of infarct progression rate in the ESCAPE-NA1 trial. J Neurointerv Surg. 2022 Sep;14(9):886-891. doi: 10.1136/neurintsurg-2021-017994. Epub 2021 Sep 7. PMID 34493575
- [Background] Olivot JM, Mlynash M, Inoue M, Marks MP, Wheeler HM, Kemp S, Straka M, Zaharchuk G, Bammer R, Lansberg MG, Albers GW; DEFUSE 2 Investigators. Hypoperfusion intensity ratio predicts infarct progression and functional outcome in the DEFUSE 2 Cohort. Stroke. 2014 Apr;45(4):1018-23. doi: 10.1161/STROKEAHA.113.003857. Epub 2014 Mar 4. PMID 24595591
- [Background] Lyden P, Buchan A, Boltze J, Fisher M; STAIR XI Consortium*. Top Priorities for Cerebroprotective Studies-A Paradigm Shift: Report From STAIR XI. Stroke. 2021 Aug;52(9):3063-3071. doi: 10.1161/STROKEAHA.121.034947. Epub 2021 Jul 22. PMID 34289707
- [Background] Nie X, Leng X, Miao Z, Fisher M, Liu L. Clinically Ineffective Reperfusion After Endovascular Therapy in Acute Ischemic Stroke. Stroke. 2023 Mar;54(3):873-881. doi: 10.1161/STROKEAHA.122.038466. Epub 2022 Dec 7. PMID 36475464
- [Background] Tiedt S, Duering M, Barro C, Kaya AG, Boeck J, Bode FJ, Klein M, Dorn F, Gesierich B, Kellert L, Ertl-Wagner B, Goertler MW, Petzold GC, Kuhle J, Wollenweber FA, Peters N, Dichgans M. Serum neurofilament light: A biomarker of neuroaxonal injury after ischemic stroke. Neurology. 2018 Oct 2;91(14):e1338-e1347. doi: 10.1212/WNL.0000000000006282. Epub 2018 Sep 14. PMID 30217937
- [Background] Anand N, Stead LG. Neuron-specific enolase as a marker for acute ischemic stroke: a systematic review. Cerebrovasc Dis. 2005;20(4):213-9. doi: 10.1159/000087701. Epub 2005 Aug 22. PMID 16123539
- [Background] Herrmann M, Vos P, Wunderlich MT, de Bruijn CH, Lamers KJ. Release of glial tissue-specific proteins after acute stroke: A comparative analysis of serum concentrations of protein S-100B and glial fibrillary acidic protein. Stroke. 2000 Nov;31(11):2670-7. doi: 10.1161/01.str.31.11.2670. PMID 11062293
- [Background] Wunderlich MT, Wallesch CW, Goertler M. Release of glial fibrillary acidic protein is related to the neurovascular status in acute ischemic stroke. Eur J Neurol. 2006 Oct;13(10):1118-23. doi: 10.1111/j.1468-1331.2006.01435.x. PMID 16987165
- [Background] Foerch C, Singer OC, Neumann-Haefelin T, du Mesnil de Rochemont R, Steinmetz H, Sitzer M. Evaluation of serum S100B as a surrogate marker for long-term outcome and infarct volume in acute middle cerebral artery infarction. Arch Neurol. 2005 Jul;62(7):1130-4. doi: 10.1001/archneur.62.7.1130. PMID 16009772
- [Background] 18. Vlegels N, Gonzalez-Ortiz F, Knuth NL, et al. Brain-derived Tau for Monitoring Brain Injury in Acute Ischemic Stroke. Under review.
- [Background] Barber PA, Demchuk AM, Zhang J, Buchan AM. Validity and reliability of a quantitative computed tomography score in predicting outcome of hyperacute stroke before thrombolytic therapy. ASPECTS Study Group. Alberta Stroke Programme Early CT Score. Lancet. 2000 May 13;355(9216):1670-4. doi: 10.1016/s0140-6736(00)02237-6. PMID 10905241
- [Background] Hacke W, Kaste M, Fieschi C, Toni D, Lesaffre E, von Kummer R, Boysen G, Bluhmki E, Hoxter G, Mahagne MH, et al. Intravenous thrombolysis with recombinant tissue plasminogen activator for acute hemispheric stroke. The European Cooperative Acute Stroke Study (ECASS). JAMA. 1995 Oct 4;274(13):1017-25. PMID 7563451
- [Background] Gonzalez-Ortiz F, Turton M, Kac PR, Smirnov D, Premi E, Ghidoni R, Benussi L, Cantoni V, Saraceno C, Rivolta J, Ashton NJ, Borroni B, Galasko D, Harrison P, Zetterberg H, Blennow K, Karikari TK. Brain-derived tau: a novel blood-based biomarker for Alzheimer's disease-type neurodegeneration. Brain. 2023 Mar 1;146(3):1152-1165. doi: 10.1093/brain/awac407. PMID 36572122
- [Background] Puetz V, Sylaja PN, Coutts SB, Hill MD, Dzialowski I, Mueller P, Becker U, Urban G, O'Reilly C, Barber PA, Sharma P, Goyal M, Gahn G, von Kummer R, Demchuk AM. Extent of hypoattenuation on CT angiography source images predicts functional outcome in patients with basilar artery occlusion. Stroke. 2008 Sep;39(9):2485-90. doi: 10.1161/STROKEAHA.107.511162. Epub 2008 Jul 10. PMID 18617663
- [Background] Austein F, Riedel C, Kerby T, Meyne J, Binder A, Lindner T, Huhndorf M, Wodarg F, Jansen O. Comparison of Perfusion CT Software to Predict the Final Infarct Volume After Thrombectomy. Stroke. 2016 Sep;47(9):2311-7. doi: 10.1161/STROKEAHA.116.013147. Epub 2016 Aug 9. PMID 27507864
- [Background] Tan IY, Demchuk AM, Hopyan J, Zhang L, Gladstone D, Wong K, Martin M, Symons SP, Fox AJ, Aviv RI. CT angiography clot burden score and collateral score: correlation with clinical and radiologic outcomes in acute middle cerebral artery infarct. AJNR Am J Neuroradiol. 2009 Mar;30(3):525-31. doi: 10.3174/ajnr.A1408. Epub 2009 Jan 15. PMID 19147716
- [Background] Menon BK, Smith EE, Modi J, Patel SK, Bhatia R, Watson TW, Hill MD, Demchuk AM, Goyal M. Regional leptomeningeal score on CT angiography predicts clinical and imaging outcomes in patients with acute anterior circulation occlusions. AJNR Am J Neuroradiol. 2011 Oct;32(9):1640-5. doi: 10.3174/ajnr.A2564. Epub 2011 Jul 28. PMID 21799045